CLINICAL TRIAL: NCT01526889
Title: A Randomized, Active-controlled, Open-label, Multicenter proof-of Concept Study of Intravitreal LFG316 in Patients With Active Non-infectious Intermediate-, Posterior-, or Panuveitis Requiring Systemic Immunosuppressive Therapy
Brief Title: Safety,Tolerability and Efficacy of Intravitreal LFG316 in Patients With Active Non-infectious Intermediate-, posterior-or Panuveitis ,
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLFG316A2204; 2011-003254-90 (EudraCT Number)
Record Dates: First submitted 2012-02-01; First posted 2012-02-06 (Estimated); Results first posted 2018-10-31 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2018-10

CONDITIONS: Non-infectious Intermediate Uveitis; Non-infectious Posterior Uveitis; Non-infectious Panuveitis
Keywords: Non-infectious uveitis; Panuveitis; Visual acuity; Vitreous Haze; Inflammation of the uvea; inflammation of the middle, pigmented vascular structures of the eye, iris, ciliary body, choroid plexus
MeSH Terms: conditions — Panuveitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LFG316 -Intravitreal Injection (Experimental)
  Interventions: Drug: LFG316
- Conventional Therapy (Active Comparator)
  Interventions: Drug: Conventional Therapy

INTERVENTIONS:
Drug: LFG316 — LFG316 administered intravitreally (IVT)
  Arms: LFG316 -Intravitreal Injection
Drug: Conventional Therapy — Conventional Therapy administered in accordance with its prescribing info.
  Arms: Conventional Therapy

SUMMARY:
This was a multi-center, randomized, active-controlled, open-label study. Approximately 24 patients with active, non-infectious intermediate-, posterior-, or panuveitis requiring systemic immunosuppressive therapy were enrolled.

Safety, efficacy, and PK assessments occurred at scheduled visits over a 12-week period. Low-molecular-weight non-steroidal immunosuppressive medications were allowed up to the baseline day as long as the dose had not changed in the 3 weeks prior to baseline, except for corticosteroid doses for which might have changed.

Patients responding to treatment were offered up to 6 months of extended treatment. Assessments for safety included laboratory safety tests, ECGs, physical exams, ocular exams, vital signs and the monitoring of adverse events. Study participation varied from a minimum of 3 months to a maximum of 9 months.

DETAILED DESCRIPTION:
Approximately 24 patients with active non-infectious uveitis, in at least one eye, requiring intensification of systemic immunosuppressive therapy were enrolled and randomized to receive intravitreal LFG316 or conventional therapy (investigator's discretion). Only one eye (the study eye) were treated with LFG316 and the other eye (fellow eye) were treated at the investigator's discretion.Throughout the study, the fellow eye might have been treated as needed; except that certain systemic medications were prohibited. There was 1 screening and 8 scheduled visits over 85 days for a total of 9 site visits for all patients.

At Day 85, patients receiving LFG316 treatment who met the criteria for a 'responder', were offered an additional 6 months of LFG316 treatment on a PRN basis. Additional 3 scheduled visits were attended by LFG316-responder patients during the extension period. However, patients could have unscheduled visits as needed and as determined by the investigator. Safety evaluation and ocular assessments were performed throughout the study duration. Patients in the treatment extension phase, who experienced a flare post their last dose and required treatment, might have received a dose of LFG316. These patients were assessed for a response at their next PRN visit as scheduled by the investigator. Visit frequency was determined by the investigator. If they continued to respond to LFG316 therapy, they might have remained in the PRN treatment arm. They might have received up to 7 additional doses of LFG316 in the PRN period. Throughout the trial LFG316 were not administered more frequently than monthly. Patients in the extension phase, who discontinued treatment prematurely were asked to return approximately 1 month after their last dose. Low molecular weight non-steroidal immunosuppressive medications were allowed up to the baseline day as long as the dose had not changed in the 3 weeks prior to baseline, except for corticosteroid doses which might have changed.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female patients 18 years or older
* Active NIU, in at least one eye, as defined below, in patients requiring intensification of systemic immunosuppressive therapy;
* Vitreous haze at least 1+ on the scale of Nussenblatt et al 1985,or
* Chorioretinal lesions due to uveitis (chorioretinal lesions due to infectious uveitis excluded)
* Patients with a flare and at the time of the enrollment on systemic corticosteroid or non-steroidal immunosuppressants had their therapy tapered or stopped, respectively, at the time of intravitreal LFG316 administration.

Visual acuity (ETDRS method) of 20 letters (20/400 Snellen equivalent) or better in the study eye.

* For female patients, must not be pregnant or lactating and must, unless post-menopausal, use effective contraception.
* Ability to provide informed consent and comply with the protocol.

Key Exclusion Criteria:

* Uveitis so severe that, in the investigator's judgment, it was too risky to test an experimental drug
* Any biologic immunosuppressive agent given via intravitreal, intravenous or subcutaneous route within 4-12 months depending on the agent.
* History of infectious uveitis or endophthalmitis in either eye.
* History of retinal detachment
* Any intraocular surgery, intravitreal injection, periocular injection, or laser photocoagulation to the study eye within 90 days prior to dosing.
* In the study eye, cataract expected to interfere with study conduct or require surgery during the study.
* Forms of uveitis that may have spontaneously resolved

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-12-20 (Actual); Primary Completion 2017-02-16 (Actual); Study Completion 2017-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- United States (6):
  - Novartis Investigative Site, Golden, Colorado
  - Novartis Investigative Site, Marietta, Georgia
  - Novartis Investigative Site, Cambridge, Massachusetts
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Teaneck, New Jersey
  - Novartis Investigative Site, Houston, Texas
- United Kingdom (2):
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=328

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Approximately 24 patients were planned to be enrolled. A total of 25 patients were randomized (18 patients in LFG316 group and 7 patients in conventional therapy group).
Groups:
- LFG316: LFG316 administered intravitreally
- Conventional Therapy: Conventional treatment was selected by the investigator
Period: Treatment Period
Arm/Group | LFG316 | Conventional Therapy
Started | 18 | 7
Completed | 16 | 7
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0
Period: Treatment Extension Period
Arm/Group | LFG316 | Conventional Therapy
Started | 5 | 0
Completed | 4 | 0
Not Completed | 1 | 0
Not completed — Administrative problems | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAS): All patients who received study drug (LFG316 or conventional treatment) were included in the safety analysis set.
Groups:
- Total: Total of all reporting groups
Arm/Group | LFG316 | Conventional Therapy | Total
Number analyzed (Participants) | 18 | 7 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: SAS
  Years | 45.3 (14.84) | 39.1 (14.89) | 43.6 (14.81)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: SAS
  Participants
    Female | 7 | 4 | 11
    Male | 11 | 3 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Safetyanalysis set
  Participants
    Hispanic or Latino | 2 | 0 | 2
    Not Hispanic or Latino | 16 | 7 | 23
    Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: SAS
  Participants
    Caucasian | 17 | 6 | 23
    Black | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response Rate for the Individual Response Criteria - in the Study Eye
Description: Response rate as defined by:
  1. An improvement of 2 or more steps in vitreous haze (scale of 0 to 4), relative to baseline OR
  2. An improvement of 10 or more letters in visual acuity (VA), relative to baseline OR
  3. An improvement of 2 or more steps in anterior chamber cells (ACC) score (scale of 0 to 4), relative to baseline OR
  4. Absence of chorioretinal lesions as determined by the investigator
Time Frame: Day 85 (end of study)
Population: Efficacy 1 analysis set: All patients in the safety analysis set who received any study treatment (LFG316 or conventional treatment) with evaluable efficacy data for at least one efficacy endpoint(s) (ocular assessments) and with no major protocol deviations that had an impact on efficacy data.
Measure: Number; unit: Participants
Arm/Group | LFG316 | Conventional Therapy
Number analyzed (Participants) | 18 | 7
Participants
  Improvement of vitreous haze ≥2 steps (N=15,6): number analyzed (Participants) | 15 | 6
  Improvement of vitreous haze ≥2 steps (N=15,6) | 3 | 3
  Improvement of VA ≥ 10 letters (N=15,6): number analyzed (Participants) | 15 | 6
  Improvement of VA ≥ 10 letters (N=15,6) | 0 | 1
  Improvement of ACC score ≥2 steps (N=7, 1): number analyzed (Participants) | 7 | 1
  Improvement of ACC score ≥2 steps (N=7, 1) | 0 | 0
  Resolution of chorioretinal lesions (N= 3, 0): number analyzed (Participants) | 3 | 0
  Resolution of chorioretinal lesions (N= 3, 0) | 0 |

2. Primary Outcome: Number of Participants With Remission in Study Eye - Treatment Period
Description: Remission (complete response) was defined as any patient who had:
  * a vitreous haze score of 0 or 0.5 (scale of 0 to 4) in the study eye, AND
  * an anterior chamber cell score of 0 (scale of 0 to 4), AND
  * no chorioretinal lesions in the study eye, AND
  * was off all immune modulatory therapy (systemic, corticosteroids and topical), AND
  * without any worsening of uveitis during the trial.
Time Frame: Day 85 (end of study)
Population: Efficacy 1 analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | LFG316 | Conventional Therapy
Number analyzed (Participants) | 18 | 7
Participants | 2 | 0

3. Secondary Outcome: Number of Participants With Vitreous Haze Score in Study Eye - Treatment Period
Description: Vitreous haze score (based on funduscopic exam): 0, 0.5/Trace, 1+, 2+, 3+, 4+
  Vitreous haze score (scale of 0 to 4) with a score of 4 being the most hazed.
Time Frame: Day 2, 8, 15, 29, 43, 57 and, 85 (end of the study)
Population: Efficacy 1 analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | LFG316 | Conventional Therapy
Number analyzed (Participants) | 18 | 7
Participants
  Day 2: number analyzed (Participants) | 15 | 7
  Day 2: 0 | 0 | 0
  Day 2: 0.5/Trace | 2 | 1
  Day 2: 1+ | 10 | 4
  Day 2: 2+ | 1 | 1
  Day 2: 3+ | 2 | 1
  Day 2: 4+ | 0 | 0
  Day 8: number analyzed (Participants) | 6 | 1
  Day 8: 0 | 0 | 0
  Day 8: 0.5/Trace | 1 | 0
  Day 8: 1+ | 4 | 1
  Day 8: 2+ | 0 | 0
  Day 8: 3+ | 1 | 0
  Day 8: 4+ | 0 | 0
  Day 15: number analyzed (Participants) | 16 | 7
  Day 15: 0 | 2 | 1
  Day 15: 0.5/Trace | 3 | 1
  Day 15: 1+ | 6 | 4
  Day 15: 2+ | 3 | 1
  Day 15: 3+ | 0 | 0
  Day 15: 4+ | 2 | 0
  Day 29: number analyzed (Participants) | 15 | 7
  Day 29: 0 | 0 | 3
  Day 29: 0.5/Trace | 4 | 1
  Day 29: 1+ | 10 | 3
  Day 29: 2+ | 0 | 0
  Day 29: 3+ | 0 | 0
  Day 29: 4+ | 1 | 0
  Day 43: number analyzed (Participants) | 14 | 6
  Day 43: 0 | 6 | 2
  Day 43: 0.5/Trace | 1 | 3
  Day 43: 1+ | 6 | 1
  Day 43: 2+ | 0 | 0
  Day 43: 3+ | 0 | 0
  Day 43: 4+ | 1 | 0
  Day 57: number analyzed (Participants) | 14 | 7
  Day 57: 0 | 5 | 2
  Day 57: 0.5/Trace | 5 | 2
  Day 57: 1+ | 4 | 3
  Day 57: 2+ | 0 | 0
  Day 57: 3+ | 0 | 0
  Day 57: 4+ | 0 | 0
  Day 85 (end of study): number analyzed (Participants) | 15 | 6
  Day 85 (end of study): 0 | 2 | 1
  Day 85 (end of study): 0.5/Trace | 6 | 3
  Day 85 (end of study): 1+ | 3 | 2
  Day 85 (end of study): 2+ | 3 | 0
  Day 85 (end of study): 3+ | 1 | 0
  Day 85 (end of study): 4+ | 0 | 0

4. Secondary Outcome: Mean Best Corrected Visual Acuity (BCVA) in Study Eye - Treatment Period
Description: Visual acuity was measured using Early Treatment Diabetic Retinopathy Study (ETDRS) eye charts under ETDRS conditions.
  ETDRS best-corrected visual acuity was obtained in each eye separately under certified ETDRS conditions. This assessment was to be performed prior to pupil dilation. The number of letters read correctly (for each eye) was recorded.
  BCVA is based on the number of letters read correctly.
Time Frame: Day 2, 8, 15, 29, 43, 57 and, 85 (end of the study)
Population: Efficacy 1 analysis set
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | LFG316 | Conventional Therapy
Number analyzed (Participants) | 18 | 7
letters
  Day 2: number analyzed (Participants) | 15 | 7
  Day 2 | 72.5 (19.36) | 76.1 (0.7)
  Day 8: number analyzed (Participants) | 6 | 1
  Day 8 | 80.5 (11.69) | 79.0 (79)
  Day 15: number analyzed (Participants) | 16 | 7
  Day 15 | 68.8 (18.53) | 78.9 (9.10)
  Day 29: number analyzed (Participants) | 15 | 7
  Day 29 | 70.3 (19.39) | 79.6 (9.47)
  Day 43: number analyzed (Participants) | 14 | 6
  Day 43 | 65.5 (24.45) | 77.3 (9.07)
  Day 57: number analyzed (Participants) | 14 | 7
  Day 57 | 72.6 (14.79) | 80.1 (10.35)
  Day 85: number analyzed (Participants) | 15 | 6
  Day 85 | 72.1 (15.53) | 76.7 (10.25)

5. Secondary Outcome: Number of Patients With Macular Edema in Study Eye - Treatment Period
Description: Macular edema is a sign of uveitis.
Time Frame: Day 85 (end of study)
Population: Efficacy 1 analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | LFG316 | Conventional Therapy
Number analyzed (Participants) | 10 | 3
Participants
  Day 2: number analyzed (Participants) | 6 | 1
  Day 2 | 2 | 1
  Day 8: number analyzed (Participants) | 6 | 1
  Day 8 | 1 | 1
  Day 15: number analyzed (Participants) | 7 | 1
  Day 15 | 3 | 0
  Day 29: number analyzed (Participants) | 7 | 1
  Day 29 | 2 | 0
  Day 43: number analyzed (Participants) | 7 | 1
  Day 43 | 2 | 0
  Day 57: number analyzed (Participants) | 8 | 2
  Day 57 | 2 | 0
  Day 85 (end of study): number analyzed (Participants) | 8 | 3
  Day 85 (end of study) | 2 | 0

6. Secondary Outcome: Number of Patients With Chorioretinal Lesions in Study Eye - Treatment Period
Description: Chorioretinal lesions is a sign of uveitis.
Time Frame: Day 2, 8, 15, 29, 43, 57 and, 85 (end of the study)
Population: Efficacy 1 analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | LFG316 | Conventional Therapy
Number analyzed (Participants) | 10 | 3
Participants
  Day 2: number analyzed (Participants) | 6 | 1
  Day 2 | 3 | 0
  Day 8: number analyzed (Participants) | 6 | 1
  Day 8 | 2 | 0
  Day 15: number analyzed (Participants) | 7 | 1
  Day 15 | 4 | 0
  Day 29: number analyzed (Participants) | 7 | 1
  Day 29 | 5 | 0
  Day 43: number analyzed (Participants) | 7 | 1
  Day 43 | 4 | 0
  Day 57: number analyzed (Participants) | 8 | 2
  Day 57 | 5 | 1
  Day 85 (end of study): number analyzed (Participants) | 8 | 3
  Day 85 (end of study) | 4 | 1

7. Secondary Outcome: Number of Participants With Anterior Chamber Cells Score in Study Eye - Treatment Period
Description: anterior chamber cells score (ACCS) with the scores being 0 (≤ 1 cell), 0.5 (1 to 5 aqueous cells), 1 (6 to 15 aqueous cells), 2 (16 to 25 aqueous cells), 3 (26 to 50 aqueous cells), 4 (>50 aqueous cells).
Time Frame: Day 2, 8, 15, 29, 43, 57 and, 85 (end of the study)
Population: Efficacy 1 analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | LFG316 | Conventional Therapy
Number analyzed (Participants) | 10 | 3
Participants
  Day 2: number analyzed (Participants) | 7 | 1
  Day 2: 0; <1 cell | 2 | 0
  Day 2: 0.5; 1-5 cells | 4 | 1
  Day 2: 1; 6-15 cells | 1 | 0
  Day 2: 2; 16-25 cells | 0 | 0
  Day 2: 3; 26-50 cells | 0 | 0
  Day 2: 4; >50 cells | 0 | 0
  Day 8: number analyzed (Participants) | 6 | 1
  Day 8: 0; <1 cell | 2 | 0
  Day 8: 0.5; 1-5 cells | 4 | 1
  Day 8: 1; 6-15 cells | 0 | 0
  Day 8: 2; 16-25 cells | 0 | 0
  Day 8: 3; 26-50 cells | 0 | 0
  Day 8: 4; >50 cells | 0 | 0
  Day 15: number analyzed (Participants) | 8 | 1
  Day 15: 0; <1 cell | 3 | 1
  Day 15: 0.5; 1-5 cells | 4 | 0
  Day 15: 1; 6-15 cells | 1 | 0
  Day 15: 2; 16-25 cells | 0 | 0
  Day 15: 3; 26-50 cells | 0 | 0
  Day 15: 4; >50 cells | 0 | 0
  Day 29: number analyzed (Participants) | 7 | 1
  Day 29: 0; <1 cell | 2 | 1
  Day 29: 0.5; 1-5 cells | 5 | 0
  Day 29: 1; 6-15 cells | 0 | 0
  Day 29: 2; 16-25 cells | 0 | 0
  Day 29: 3; 26-50 cells | 0 | 0
  Day 29: 4; >50 cells | 0 | 0
  Day 43: number analyzed (Participants) | 7 | 1
  Day 43: 0; <1 cell | 5 | 1
  Day 43: 0.5; 1-5 cells | 0 | 0
  Day 43: 1; 6-15 cells | 1 | 0
  Day 43: 2; 16-25 cells | 1 | 0
  Day 43: 3; 26-50 cells | 0 | 0
  Day 43: 4; >50 cells | 0 | 0
  Day 57: number analyzed (Participants) | 8 | 2
  Day 57: 0; <1 cell | 5 | 1
  Day 57: 0.5; 1-5 cells | 1 | 1
  Day 57: 1; 6-15 cells | 2 | 0
  Day 57: 2; 16-25 cells | 0 | 0
  Day 57: 3; 26-50 cells | 0 | 0
  Day 57: 4; >50 cells | 0 | 0
  Day 85: number analyzed (Participants) | 9 | 3
  Day 85: 0; <1 cell | 4 | 3
  Day 85: 0.5; 1-5 cells | 5 | 0
  Day 85: 1; 6-15 cells | 0 | 0
  Day 85: 2; 16-25 cells | 0 | 0
  Day 85: 3; 26-50 cells | 0 | 0
  Day 85: 4; >50 cells | 0 | 0

8. Secondary Outcome: Number of Participants With or Without Anti-LFG316 Antibodies
Description: Blood will be collected at each visit for the profiling of serum drug concentrations. The summary of immunogenicity (IG) by visit . The immunogenicity data (presence/absence of anti-LFG316 antibodies [anti-drug antibodies]).
  NO: No immunogenicity; YES: Positive immunogenicity.
Time Frame: Throughout the study (treatment and extension period), up to day 271
Population: Pharmacokinetic analysis set: All patients in the safety analysis set with evaluable PK data and with no protocol deviations affecting PK data.
Measure: Count of Participants; unit: Participants
Arm/Group | LFG316
Number analyzed (Participants) | 17
Participants
  Day 1: number analyzed (Participants) | 15
  Day 1: participants with anti-LFG316 antibodies | 3
  Day 1: participants without anti-LFG316 antibodies | 12
  Day 29: number analyzed (Participants) | 13
  Day 29: participants with anti-LFG316 antibodies | 3
  Day 29: participants without anti-LFG316 antibodies | 10
  Day 85 (end of study): number analyzed (Participants) | 11
  Day 85 (end of study): participants with anti-LFG316 antibodies | 2
  Day 85 (end of study): participants without anti-LFG316 antibodies | 9
  Day 169: number analyzed (Participants) | 2
  Day 169: participants with anti-LFG316 antibodies | 1
  Day 169: participants without anti-LFG316 antibodies | 1
  Day 253: number analyzed (Participants) | 1
  Day 253: participants with anti-LFG316 antibodies | 0
  Day 253: participants without anti-LFG316 antibodies | 1
  End of extension period: number analyzed (Participants) | 1
  End of extension period: participants with anti-LFG316 antibodies | 1
  End of extension period: participants without anti-LFG316 antibodies | 0

9. Secondary Outcome: Mean Percent Change in Total C5 Concentrations in Serum - Treatment Period
Description: Percent change from baseline (using each patient's pre-dose value as baseline) in total C5 concentrations.
Time Frame: Day 2, 15, 29, 43, 57 and, 85 (end of the study)
Population: Pharmacodynamic (PD) analysis set: All patients in the safety analysis set with EVALUABLE pharmacodynamics (PD) data (Total C5) and with no major protocol deviations that had an impact on PD data were included in the PD analysis set.
Measure: Mean (Standard Deviation); unit: Percent change in C5
Arm/Group | LFG316 | Conventional Therapy
Number analyzed (Participants) | 15 | 7
Percent change in C5
  Day 2 | 6.80 (14.5) | 1.02 (5.69)
  Day 15: number analyzed (Participants) | 14 | 7
  Day 15 | 8.21 (15.3) | -1.27 (19.7)
  Day 29: number analyzed (Participants) | 15 | 6
  Day 29 | 10.6 (17.4) | -8.33 (17.5)
  Day 43: number analyzed (Participants) | 12 | 5
  Day 43 | 8.38 (13.4) | 6.46 (18.6)
  Day 57: number analyzed (Participants) | 15 | 5
  Day 57 | 6.73 (12.0) | 5.98 (40.9)
  Day 85: number analyzed (Participants) | 13 | 7
  Day 85 | 3.21 (22.1) | 1.28 (31.3)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 5 years.
Groups:
- LFG316: LF G316 administered intravitreally
Arm/Group | LFG316 | Conventional Therapy
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/7
Other Adverse Events (participants affected / at risk) | 11/18 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LFG316 (N=18) | Conventional Therapy (N=7)
Retinal detachment (Eye disorders) | 1 | 0
Retinopathy proliferative (Eye disorders) | 1 | 0
Mycotic endophthalmitis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LFG316 (N=18) | Conventional Therapy (N=7)
Cataract (Eye disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 4 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0
Cystoid macular oedema (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 1
Eye pain (Eye disorders) | 1 | 0
Hypotony of eye (Eye disorders) | 0 | 1
Macular fibrosis (Eye disorders) | 1 | 1
Ocular hypertension (Eye disorders) | 0 | 1
Uveitis (Eye disorders) | 4 | 0
Visual impairment (Eye disorders) | 1 | 0
Vitreous floaters (Eye disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Giardiasis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 2 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Intraocular pressure increased (Investigations) | 3 | 0
Optic nerve cup/disc ratio increased (Investigations) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT01526889/SAP_000.pdf
  • Study Protocol (2015-09-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT01526889/Prot_001.pdf